CLINICAL TRIAL: NCT01312870
Title: Prospective Randomized Study of Postoperative Nutritional Support in Cardiac Surgery.
Brief Title: Study of Postoperative Nutritional Support in Cardiac Surgery.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, Anesthesist, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNSICP-71421
Record Dates: First submitted 2011-03-02; First posted 2011-03-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- postoperative nutritional supplements (Experimental): postoperative nutritional supplements in addition to standard hospital diet
  Interventions: Dietary Supplement: Ensure, Abbott Nutrition
- standard hospital diet (Placebo Comparator): patients receiving standard hospital diet
  Interventions: Other: standard hospital diet

INTERVENTIONS:
Dietary Supplement: Ensure, Abbott Nutrition — Enteral feeding Ensure, Abbott Nutrition 400 ml per day for seven postoperative days
  Arms: postoperative nutritional supplements
Other: standard hospital diet — standard hospital diet
  Arms: standard hospital diet

SUMMARY:
The purpose of this study is to determine whether postoperative nutritional support improves postoperative outcomes in cardiac patients with malnutrition .

ELIGIBILITY:
Inclusion Criteria:

* Absolute lymphocyte count < 1500
* Albumin <35 g/L
* Body mass index<21 kg/m2
* "B" class of nutritional status according to Subjective Global Assessment

Exclusion Criteria:

* Hepatitis B, C
* Total circulatory arrest
* Absence of informed consent signed
* Chronic liver diseases
* Gastric resection in patient's history
* Physical limitations of normal feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 month

SECONDARY OUTCOMES:
Postoperative complications | 1 month
  Cardiac arrhythmia, infectious complications.
Total lymphocyte count | before operation, 7, 14, 21 postoperative days
Serum albumin | Before operation, 7, 14, 21 postoperaitve days
Serum prealbumin | Before operation, 7, 14, 21 postoperaitve days
Retinol-binding protein | Before operation, 7, 14, 21 postoperaitve days

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk
  - State Research Institute of CIrculation Pathology, Novosibirsk